CLINICAL TRIAL: NCT05424991
Title: The Effect of Comedy Film on Preoperative Anxiety and Postoperative Pain Level in Abdominal Surgery Patients
Brief Title: The Effect of Comedy Film on Preoperative Anxiety and Postoperative Pain Level.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gurkan KAPIKIRAN (Other)
Responsible Party: Sponsor-Investigator, Gurkan KAPIKIRAN, Assistant Professor, Malatya Turgut Ozal University
Organization: Malatya Turgut Ozal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021/179
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: General Surgery; Anxiety; Pain
Keywords: Abdominal Surgery; Preoperative Anxiety; Comedy Film; Postoperative Pain
MeSH Terms: conditions — Anxiety Disorders; Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comedy movie group (Experimental): The anxiety level of the patients in the experimental group was measured. Afterwards, each patient watched a comedy movie for 25 minutes. Anxiety levels were re-measured 25 minutes after watching the comedy movie. Pain levels were measured after the anesthesia effect disappeared in the postoperative period. Afterwards, each patient watched a comedy movie for 25 minutes. Pain levels were re-measured 25 minutes after watching the comedy movie.
  Interventions: Behavioral: comedy movie group
- No treatment group (No Intervention): In the follow-up of the patient, no application was made other than clinical protocols. Anxiety scale was filled preoperatively, and anxiety level was evaluated again 25 minutes later. Pain level was evaluated in the postoperative period. Pain levels were evaluated again at the end of the same period with the experimental group without any intervention.

INTERVENTIONS:
Behavioral: comedy movie group — The patients watched the collage videos of Turkish cinema Yeşilçam comedy films created by the researchers for 25 minutes. The videos were created by making collages from videos on youtube.
  Arms: comedy movie group

SUMMARY:
When we look at the literature, studies examining the effect of having patients watch comedy films on anxiety and pain are limited. However, it was observed that the anxiety and pain levels of oncology patients who underwent surgery decreased by watching comedy movies. Therefore, in order to use the healing effects of humor, our study was planned to determine the effect of watching comedy films on the level of anxiety and postoperative pain in patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Whether it is major surgery or minor surgery, preoperative anxiety is observed in all patients in the preoperative period. A high level of anxiety causes many physiological and psychological problems in the body and causes an increase in sympathetic and endocrine system stimuli. Among the physiological and psychological problems seen, many conditions such as recovery time, quality of life, health care expenditures, vital signs and well-being are negatively affected. Therefore, many applications can be used to reduce the level of anxiety before surgery. With humor, which is one of them, the anxiety levels of the patients can be reduced and they can manage their stress management better. In addition to reducing the level of anxiety before the operation, the experience of post-operative pain is one of the important problems experienced by the patients. Pain complaints are a general problem in the postoperative period in abdominal surgeries. The usefulness of using supportive complementary and alternative therapies in addition to pharmacological treatments in postoperative pain management is emphasized in the literature. Among these non-pharmacological treatments, it is stated that humor and laughter increase tolerance to pain and have positive effects on mood. Humor and laughter not only increase pain tolerance, but also reduce fear, anxiety and anger, and help lower the level of anxiety. Therefore, in order to use the healing effects of humor, our study was planned to determine the effect of watching comedy films on the level of anxiety and postoperative pain in patients undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Defining the postoperative pain intensity of 4 and above,
* No cognitive problem
* Willing to participate in the research
* Having had Abdominal Surgery.

Exclusion Criteria:

* with a communication barrier,
* Having an uncontrollable psychiatric disorder,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Pain level | Time Frame: 0-20 minutes
  It is a measure of pain level. Pain intensity ranges from 0 to 10, 0 points no pain, 10 points unbearable pain.
Anxiety Level | 0-20 minutes
  The state anxiety scale is a 4-point Likert type measurement tool consisting of 20 questions. The items of the scale that are positive and increase the total anxiety score; Items 3, 4, 6, 7, 9, 12, 13, 14, 17, 18. The items of the scale that are negative and decrease the total anxiety level; Articles 1, 2, 5, 8, 10, 11, 15, 16, 19, 20. While evaluating, positive items are calculated as 1,2,3,4 points. Negative items are calculated as -1, -2, -3, -4 points. A 50 point constant is added to the obtained scores, and an average score between 20-80 points is obtained. The higher the total anxiety score, the higher the anxiety level.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers can reach and get information by e-mail.